CLINICAL TRIAL: NCT03356093
Title: Change in Symptom Clusters in HNC Patients Undergoing Postoperative Radiotherapy: A Longitudinal Study
Brief Title: Change in Symptom Clusters in HNC Patients
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Chia-Chin Lin, Head and Professor, Taipei Medical University
Other Study IDs: HKU_2
Record Dates: First submitted 2017-11-20; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Head and Neck
Keywords: head and neck cancer, symptom cluster, change, radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with head and neck cancer: No intervention was provided. The patients were only asked to complete a set of questionnaire at baseline, and week 1, 2, 3, 4, 5 and 6 after starting of postoperative radiotherapy.
  Interventions: Other: complete questionnaire

INTERVENTIONS:
Other: complete questionnaire — Patients were asked to complete a questionnaire at baseline, and week 1, 2, 3, 4, 5 and 6 after starting of radiotherapy.

SUMMARY:
Head and neck cancer (HNC) is the sixth most common malignancy worldwide, causing more than 379,000 deaths in 2015 notwithstanding the breakthrough in cancer screening and medical treatment. The primary treatment for HNC is a combination of surgery and radiotherapy, either delivered preoperatively or postoperatively. Although these treatments, especially the postoperative radiotherapy can greatly improve the survival of patients, they still have to pay a high price for numerous symptoms induced by radiation. On the other hand, research on symptoms clusters is an emerging field in oncology which aims to understand the complexity of multiple symptoms experienced by cancer patients. A thorough understanding of symptom clusters help informs the development of comprehensive care plans which target a group of symptoms that is likely to coexist, thus easing the total symptom burden in cancer patients.To date, there has been a paucity of evidence regarding symptom clusters of HNC. To address the gap in existing literature, this study described the symptom clusters among HNC patients who were treated with surgery with a combination of postoperative radiotherapy. In addition, a longitudinal approach was employed to examine the change in symptom clusters throughout the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with HNC,
* Aged older than 18 years,
* Without receiving any radiotherapy prior to surgery,
* No cognitive impairment and able to communicate in Mandarin or Taiwanese

Exclusion Criteria:

- Undergoing any concurrent treatment for cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head and neck cancer patients undergoing postoperative radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | 6 months after radiotherapy
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.

SECONDARY OUTCOMES:
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | baseline
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | 1 month after radiotherapy
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | 2 months after radiotherapy
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | 3 months after radiotherapy
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | 4 months after radiotherapy
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.
treatment-related symptoms of head and neck cancer patients with post-operative radiotherapy assessed by the Taiwanese version of the MD Anderson Symptom Inventory | 5 months after radiotherapy
  The Taiwanese version of the MD Anderson Symptom Inventory is designed to assess the severity of 13 symptoms that are most commonly reported by patients undergoing cancer treatment. The symptoms include dry mouth, fatigue, sleep disturbance, pain, drowsiness, lack of appetite, nausea, vomiting, shortness of breath, numbness, difficulty remembering, distress and sadness. Participants in this study were asked to rate the severity of these symptoms on a 11-point Likert scale, with "0" representing "not present "and "10" representing "as bad as you can imagine". The item scores of 1 - 4, 5 - 6 and 7 - 10 are considered as mild, moderate and severe, respectively. The composite score can be obtained by averaging the 13 item scores.

IPD SHARING:
Plan to Share IPD: No